CLINICAL TRIAL: NCT04967417
Title: Pembrolizumab With Standard Cytotoxic Chemotherapy in Treatment Naive Non-small Cell Lung Cancer Patients With Asymptomatic Brain Metastases
Brief Title: Pembrolizumab With Standard Cytotoxic Chemotherapy in Treatment Naive NSCLC Patients With Asymptomatic Brain Metastases
Acronym: PHOEBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Clinical Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-06-008
Record Dates: First submitted 2021-06-29; First posted 2021-07-19 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; pembrolizumab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Non-squamous cell carcinoma:
  4 cycles of pemetrexed 500mg/m2 + carboplatin AUC 5.0 + pembrolizumab 200mg every 3 weeks Followed by pemetrexed 500mg/m2 + pembrolizumab 200mg every 3 weeks up to 35 cycles
  Squamous cell carcinoma:
  4 cycles of paclitaxel 200mg/m2 + carboplatin AUC 6.0 + pembrolizumab 200mg every 3 weeks Followed by pembrolizumab 200mg every 3 weeks up to 35 cycles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-squamous cell carcinoma (Experimental): * 4 cycles of pemetrexed 500mg/m2 + carboplatin AUC 5.0 + pembrolizumab 200mg every 3 weeks
  * Followed by pemetrexed 500mg/m2 + pembrolizumab 200mg every 3 weeks up to 35 cycles
  Interventions: Drug: Pemetrexed, Carboplatin, Pembrolizumab
- Squamous cell carcinoma (Experimental): * 4 cycles of paclitaxel 200mg/m2 + carboplatin AUC 6.0 + pembrolizumab 200mg every 3 weeks
  * Followed by pembrolizumab 200mg every 3 weeks up to 35 cycles
  Interventions: Drug: Paclitaxel, Carboplatin, Pembrolizumab

INTERVENTIONS:
Drug: Pemetrexed, Carboplatin, Pembrolizumab — * Pemetrexed 500mg/m2
  * Carboplatin AUC 5.0
  * Pembrolizumab 200mg
  Other Names: Alimta, Preizer carboplatin, keytruda
  Arms: Non-squamous cell carcinoma
Drug: Paclitaxel, Carboplatin, Pembrolizumab — * Paclitaxel 200mg/m2
  * Caboplatin AUC 6.0
  * Pembrolizumab 200mg
  Other Names: Anzatax, Preizer carboplatin, keytruda
  Arms: Squamous cell carcinoma

SUMMARY:
This is a Phase II single center, open-label, single arm study in patients with advanced non-small cell lung cancer (stage IV) with brain metastases.

This study will be treated with combination of Pembrolizumab 200mg plus platinum doublet based on histology subtypes.

DETAILED DESCRIPTION:
This is a Phase II single center, open-label, single arm study in patients with advanced non-small cell lung cancer (stage IV) with brain metastases. Patients will be treated with combination of Pembrolizumab 200mg plus platinum doublet based on histology subtypes. After the 4 cycles of combination phase with cytotoxic chemotherapy, maintenance phase will be followed for maximum of 35 cycles. If the disease progression is observed in CNS only which can be controlled with local treatment, systemic treatment can be continued as beyond disease progression.

Non-squamous cell carcinoma:

4 cycles of pemetrexed 500mg/m2 + carboplatin AUC 5.0 + pembrolizumab 200mg every 3 weeks Followed by pemetrexed 500mg/m2 + pembrolizumab 200mg every 3 weeks up to 35 cycles

Squamous cell carcinoma:

4 cycles of paclitaxel 200mg/m2 + carboplatin AUC 6.0 + pembrolizumab 200mg every 3 weeks Followed by pembrolizumab 200mg every 3 weeks up to 35 cycles

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 19 years of age on the day of signing informed consent with histologically confirmed diagnosis of stage IV non-small cell lung cancer with brain metastases will be enrolled in this study.
2. Must have at least one intracranial target lesion. Intracranial lesion must be equal or greater than the 10mm in longest diameter.
3. Have confirmation that EGFR or ALK-directed therapy is not indicated
4. Have measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Otherwise, previously treated with radiation is not considered as measurable lesion.
5. Have not received prior systemic treatment for their advanced/metastatic NSCLC. Subjects who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the development of metastatic disease.
6. Have a life expectancy of at least 3 months
7. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
8. Have adequate organ function
9. Male participants: A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
10. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
    * b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
11. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to IP administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents prior to IP administration as a metastatic disease treatment, including tyrosine kinase inhibitor.
4. Had major surgery < 3 weeks prior to first dose
5. No measurable CNS lesion other than CNS lesion treated with stereotactic radiotherapy or surgery
6. Had received whole brain radiotherapy or stereotactic radiotherapy to CNS disease.
7. Has received prior radiotherapy within 1 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation to non-CNS disease.
8. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
9. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, thyroid cancer or early gastric cancer or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
12. Has known active carcinomatous meningitis.
13. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
15. Has a history of (non-infectious) pneumonitis that currently required steroids or has current pneumonitis.
16. Has an active infection requiring systemic therapy.
17. Has a known history of Human Immunodeficiency Virus (HIV) infection.
18. Has a active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive with HBV DNA positive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. These patients can be participated with appropriate treatment and prophylactic treatment based on the investigator's decision.
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
22. Has had an allogenic tissue/solid organ transplant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, MD, phD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnamgu, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-squamous Cell Carcinoma: * 4 cycles of pemetrexed 500mg/m2 + carboplatin AUC 5.0 + pembrolizumab 200mg every 3 weeks
  * Followed by pemetrexed 500mg/m2 + pembrolizumab 200mg every 3 weeks up to 35 cycles
  Pemetrexed, Carboplatin, Pembrolizumab: - Pemetrexed 500mg/m2
  * Carboplatin AUC 5.0
  * Pembrolizumab 200mg
- Squamous Cell Carcinoma: * 4 cycles of paclitaxel 200mg/m2 + carboplatin AUC 6.0 + pembrolizumab 200mg every 3 weeks
  * Followed by pembrolizumab 200mg every 3 weeks up to 35 cycles
  Paclitaxel, Carboplatin, Pembrolizumab: - Paclitaxel 200mg/m2
  * Caboplatin AUC 6.0
  * Pembrolizumab 200mg
Period: Overall Study
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Started | 11 | 2
Completed | 8 | 2
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma | Total
Number analyzed (Participants) | 11 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.75) | 49 (24.04) | 61.69 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 11 | 2 | 13
Smoking history [Count of Participants; unit: Participants]
  Never | 6 | 1 | 7
  Former | 4 | 1 | 5
  Current | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Objective Response Rate
Description: Intracranial objective response is defined as the investigator's best non-confirmed response as CR (complete response) or PR (partial response) as determined using RECIST v1.1. Subjects who do not meet these criteria, including those without a post-baseline tumor assessment, are considered non-responders. Intracranial objective response rate (iORR) is defined as the proportion of subjects who achieved an objective response among all subjects treated with the IP who had measurable disease at baseline.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of t the diameters of target lesion.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 11 | 2
Participants
  Partial Response | 6 | 0
  Stable Response | 5 | 0
  Progressive Disease | 0 | 1
  Not evaluabe | 0 | 1

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the period between the start date of the investigational drug and the date of the first documented disease progression or death, whichever occurs first.
  - PFS (month) = (date of the first documented disease progression or death - date of the start of the investigational drug + 1) / 30.4375
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of diameters of TLs, taking as reference the smallest sum of diameters (nadir) on study (this includes the baseline sum if that is the smallest on study), or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: The time until the date of either disease progression or the all-cause mortality from the date of IP administration. Up to 30 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 11 | 2
Months | 7.23 [2.4 to 12.29] | 7.7 [1.25 to 14.16]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined by date of all-cause mortality from the date of IP Administration will be calculated.
Time Frame: The time until defined by date of all-cause mortality from the date of IP Administration. Up to 30 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 11 | 2
Months | 10.45 [7.2 to 21.52] | 12.45 [10.71 to 14.19]

4. Secondary Outcome: Intracranial Duration of Response
Description: The duration for intracranial response will be calculated separately to evaluate the intracranial efficacy of IP drug
Time Frame: Up to 30 months.
Population: For squamous cell carcinoma (SCC), there was no response in a total of 2 patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 11 | 0
Months | 9.3 [3.98 to 20.34] |

5. Secondary Outcome: Intracranial Progression-free Survival
Description: Progression free survival of intracranial disease defined by the date of disease progression of intracranial lesion from the date of IP administration will be calculated.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of diameters of TLs, taking as reference the smallest sum of diameters (nadir) on study (this includes the baseline sum if that is the smallest on study), or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 30 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 11 | 2
Months | 9.82 [5.19 to 21.49] | 7.7 [1.25 to 14.16]

6. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as the investigator's best non-confirmed response as CR (complete response) or PR (partial response) as determined using RECIST v1.1. Subjects who do not meet these criteria, including those without a post-baseline tumor assessment, are considered non-responders. objective response rate (ORR) is defined as the proportion of subjects who achieved an objective response among all subjects treated with the IP who had measurable disease at baseline.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of t the diameters of target lesion.
Time Frame: Up to 30 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 11 | 2
Participants
  Partial Response | 6 | 0
  Stable Disease | 4 | 0
  Progressive Disease | 1 | 1
  Not evaluable | 0 | 1

7. Secondary Outcome: Adverse Events
Description: Adverse event will be evaluated using CTCAE v5.0
Time Frame: from the date of informed consent signature to 30 days after last drug administration
Measure: Number; unit: Number
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 11 | 2
Number
  TEAEs | 11 | 2
  ADR | 5 | 0
  SAE | 2 | 0

8. Other Pre Specified Outcome: Exploratory Analyses Based on PD-L1 Expression
Description: The exploratory analyses based on the PD-L1 expression (by DAKO PD-L1 22C3 assay) from the baseline samples will be used for the exploratory analyses in subjects who are available for the PD-L1 test
Time Frame: Up to 30 months.
Population: Although this outcome was pre-specified, the study enrolled only 13 participants and valid PD-L1 expression data were available for very few participants. As such, it was not possible to conduct any meaningful exploratory analyses based on PD-L1 status. Given the limited sample size and incomplete biomarker data, this outcome was not analyzed, and no results are reported.
  All samples were collected and handled in accordance with participants' ICF and the protocol approved by the IRB.
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 28 days (±7 days) after the final administration of the study drug, up to 24months. All-Cause Mortality was assessed through study completion, up to 30 months
Arm/Group | Non-squamous Cell Carcinoma | Squamous Cell Carcinoma
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/2
Other Adverse Events (participants affected / at risk) | 11/11 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-squamous Cell Carcinoma (N=11) | Squamous Cell Carcinoma (N=2)
ALT Increased (Infections and infestations) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
AST increased (Infections and infestations) | 1 (1) | 0 (0)
AV block complete (Cardiac disorders) | 1 (1) | 0 (0)
Acute pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Aspiration pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-squamous Cell Carcinoma (N=11) | Squamous Cell Carcinoma (N=2)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute Investigations (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Infections and infestations) | 11 (11) | 0 (0)
Aspartate aminotransferase increased (Infections and infestations) | 9 (9) | 0 (0)
Blood alkaline phosphatase increased (Infections and infestations) | 2 (2) | 0 (0)
Blood bilirubin increased (Infections and infestations) | 1 (1) | 0 (0)
Blood creatine increased (Infections and infestations) | 3 (3) | 0 (0)
Weight decreased (Infections and infestations) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT04967417/Prot_000.pdf